CLINICAL TRIAL: NCT00204022
Title: A Randomized Multicenter Trial Comparing Mycophenolate Mofetil and Azathioprine as Remission-maintaining Treatment for Proliferative Lupus Glomerulonephritis. The MAINTAIN Nephritis Trial.
Brief Title: Mycophenolate Mofetil Versus Azathioprine for Maintenance Therapy of Lupus Nephritis.
Acronym: MAINTAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Frédéric A. Houssiau, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Frédéric A. Houssiau, MD, PhD, Professeur Ordinaire, Chef de Service Clinique, Université Catholique de Louvain
Organization: Université Catholique de Louvain (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EWPSLE-LN-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Lupus Nephritis
Keywords: Lupus nephritis; Treatment; Maintenance therapy; Mycophenolate mofetil; Azathioprine
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Mycophenolate mofetil (target dose 2g/day)
  Interventions: Drug: Mycophenolate mofetil
- 2 (Active Comparator): Azathioprine (target dose 2mg/kg/day)
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Mycophenolate mofetil — Mycophenolate mofetil
  Arms: 1
Drug: Azathioprine — Azathioprine
  Arms: 2

SUMMARY:
The purpose of the study is to determine whether mycophenolate mofetil is superior to azathioprine to prevent flares of lupus nephritis.

DETAILED DESCRIPTION:
Proliferative glomerulonephritis is a common and severe manifestation of systemic lupus erythematosus (SLE) that usually requires intensive therapy with high doses of glucocorticosteroids and cytotoxic drugs, such as intravenous (IV) cyclophosphamide (CYC). The objective of the MAINTAIN Nephritis Trial is to compare mycophenolate mofetil (MMF) and azathioprine (AZA), in terms of efficacy and toxicity, as remission-maintaining treatment of proliferative lupus glomerulonephritis, after a remission-inducing therapy with a short-course IV CYC regimen. The hypothesis addressed by the MAINTAIN Nephritis Trial is that MMF is superior to AZA.

ELIGIBILITY:
Inclusion Criteria:

* SLE aged ≥ 14 years
* Proteinuria ≥ 500 mg/day
* Biopsy-proven proliferative lupus nephritis

Exclusion Criteria:

* Recent treatment with high-dose glucocorticoids
* Recent treatment with immunosuppressive drugs
* More exclusion criteria in the protocol

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2001-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Time to renal flare | 5 years

SECONDARY OUTCOMES:
Number of withdrawals due to toxicity | 5 years and 10 years
Cumulated glucocorticoid intake | 5 years and 10 years
Number of treatment failures | 5 years and 10 years
24-hour proteinuria over time | 5 years and 10 years
Serum creatinine titers | 5 years and 10 years
Time to renal flare | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric A Houssiau, MD, PhD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Université catholique de Louvain, Brussels, Belgium

REFERENCES:
- [Derived] Tamirou F, Lauwerys BR, Dall'Era M, Mackay M, Rovin B, Cervera R, Houssiau FA; MAINTAIN Nephritis Trial Investigators. A proteinuria cut-off level of 0.7 g/day after 12 months of treatment best predicts long-term renal outcome in lupus nephritis: data from the MAINTAIN Nephritis Trial. Lupus Sci Med. 2015 Nov 12;2(1):e000123. doi: 10.1136/lupus-2015-000123. eCollection 2015. PMID 26629352
- [Derived] Tamirou F, D'Cruz D, Sangle S, Remy P, Vasconcelos C, Fiehn C, Ayala Guttierez Mdel M, Gilboe IM, Tektonidou M, Blockmans D, Ravelingien I, le Guern V, Depresseux G, Guillevin L, Cervera R, Houssiau FA; MAINTAIN Nephritis Trial Group. Long-term follow-up of the MAINTAIN Nephritis Trial, comparing azathioprine and mycophenolate mofetil as maintenance therapy of lupus nephritis. Ann Rheum Dis. 2016 Mar;75(3):526-31. doi: 10.1136/annrheumdis-2014-206897. Epub 2015 Mar 10. PMID 25757867